CLINICAL TRIAL: NCT03155139
Title: Primary Aldosteronism In Hypertensive Patients in China
Acronym: PA-China
Status: Completed | Type: Observational
Sponsor: Qifu Li (Other)
Collaborators: Fu Wai Hospital, Beijing, China (Other)
Responsible Party: Sponsor-Investigator, Qifu Li, Primary Investigator, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Other Study IDs: PA-China 2017
Record Dates: First submitted 2017-04-28; First posted 2017-05-16 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Hyperaldosteronism; Primary; Hypertension Secondary
Keywords: prevalence; primary aldosteronism; hypertension; nationwide
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Some subtye of PA such as glucocorticoid remediable aldosteronism(GRA) should be diagnosed by DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without primary aldosteronism (PA): PA case detection or confirmatory tests was negative.
  Interventions: Diagnostic Test: Aldosterone/renin ratio (ARR) testing
- Patients with primary aldosteronism (PA): PA case detection and confirmatory tests were positive.
  Interventions: Diagnostic Test: Aldosterone/renin ratio (ARR) testing; Diagnostic Test: Confirmatory tests

INTERVENTIONS:
Diagnostic Test: Aldosterone/renin ratio (ARR) testing — Plasma aldosterone concentration tests, Direct renin concentration tests
Diagnostic Test: Confirmatory tests — Captopril challenge test, Saline infusion test
  Groups: Patients with primary aldosteronism (PA)

SUMMARY:
To investigate the prevalence of primary aldosteronism (PA) in Chinese patients with newly diagnosed hypertension.

DETAILED DESCRIPTION:
This is a nationwide sampling study. To investigate the prevalence of primary aldosteronism (PA) in Chinese patients with hypertension, we will conduct a case detection of PA in Chinese hypertensive patients from 10 centers of China (including Beijing, Chongqing, Shanghai, Guangzhou, et al.); furthermore, a case confirmation of PA (captopril challenge test and saline infusion test) will be performed if the result of case detection is positive. This study will be completed in two years.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed hypertension(with a course less than six months);
2. Drug negative, or voluntary to discontinue/change the anti-hypertensive medications;
3. Aged between 18-80 year, gender is not limited;
4. Voluntary to sign on the informed consent.

Exclusion Criteria:

1. patients with severe cardiac, hepatic or renal dysfunction;
2. suspicious or confirmed other types of secondary hypertension, including Cushing's syndrome, pheochromocytoma and renal artery stenosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sampling Design: hypertensive patients will be continuously sampled for case detection in each center. PASS 11.0 Software-Confidence Intervals for One Proportion was used to calculate the sample size. A sample size of 2928 produces a two-sided 95% confidence interval with a width equal to 0.02 when the sample proportion(prevalence of PA) is 0.080. Accounting for the 20% withdraw rate in the process of case detection, the final sample size should be 3635 (about 4000 cases).
Sampling Method: Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2017-06-03 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects with newly diagnosed hypertension | 2 years
  To calculate the prevalence of PA in Chinese patients with hypertension
Number of subjects with confirmed primary aldosteronism (PA) | 2 years
  To calculate the prevalence of PA in Chinese patients with hypertension
Prevalence of PA | 2 years
  Prevalence of PA= Number of PA / Number of subjects with hypertension

SECONDARY OUTCOMES:
Age | 2 years
  Characteristics of PA in Chinese patients with hypertension
Blood pressure | 2 years
  Characteristics of PA in Chinese patients with hypertension
Family history of hypertension | 2 years
  Characteristics of PA in Chinese patients with hypertension
Fasting blood glucose | 2 years
  Characteristics of PA in Chinese patients with hypertension
Cardiovascular events | 2 years
  Characteristics of PA in Chinese patients with hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cai, phD, Principal Investigator — Hypertension Center, Fuwai Hospital, State Key Laboratory of Cardiovascular Disease of China
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li X, Goswami R, Yang S, Li Q. Aldosterone/direct renin concentration ratio as a screening test for primary aldosteronism: A meta-analysis. J Renin Angiotensin Aldosterone Syst. 2016 Aug 17;17(3):1470320316657450. doi: 10.1177/1470320316657450. Print 2016 Jul. PMID 27534428
- [Result] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Result] Kayser SC, Dekkers T, Groenewoud HJ, van der Wilt GJ, Carel Bakx J, van der Wel MC, Hermus AR, Lenders JW, Deinum J. Study Heterogeneity and Estimation of Prevalence of Primary Aldosteronism: A Systematic Review and Meta-Regression Analysis. J Clin Endocrinol Metab. 2016 Jul;101(7):2826-35. doi: 10.1210/jc.2016-1472. Epub 2016 May 12. PMID 27172433
- [Derived] Xu Z, Yang J, Hu J, Song Y, He W, Luo T, Cheng Q, Ma L, Luo R, Fuller PJ, Cai J, Li Q, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Primary Aldosteronism in Patients in China With Recently Detected Hypertension. J Am Coll Cardiol. 2020 Apr 28;75(16):1913-1922. doi: 10.1016/j.jacc.2020.02.052. PMID 32327102